CLINICAL TRIAL: NCT06633211
Title: Clinical and Histological Effects of the Adjunctive Use of Polynucleotide and Hyaluronic Acid-based Gel in Alveolar Preservation After Tooth Extraction: A Randomized Clinical Trial
Brief Title: Adjunctive Use of Polynucleotide and Hyaluronic Acid-based Gel in Alveolar Preservation After Tooth Extraction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adrià Jorba García (Other)
Responsible Party: Sponsor-Investigator, Adrià Jorba García, DDS, MS, University of Barcelona
Organization: University of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Regenfast
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Bone Substitutes; Tooth Extraction Status Nos
Keywords: Alveolar Ridge preservation; Guided bone regeneration

STUDY DESIGN:
Intervention Model Description: Two parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the interventional nature of the study, the surgeon cannot be blinded. A randomization sequence will be generated, and each patient will be assigned a number. To ensure allocation concealment, the surgeon will be blinded to the group assignment of each patient until just before performing the alveolar preservation procedure. The investigator responsible for conducting the radiological measurements and the histomorphometric study will be blinded to the patient's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBBM + collagen matrix (Active Comparator): An alveolar ridge preservation will be performed using particulate xenograft DBBM (Bio-Oss, Geistlich Pharma AG, Wolhusen, Switzerland), and the alveolus will be sealed with a collagen matrix (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switzerland).
  Interventions: Procedure: Alveolar ridge preservation using DBBM + collagen matrix
- DBBM + Regenfast + collagen matrix (Experimental): An alveolar preservation will be performed by means of a particulate DBBM xenograft (Bio-Oss, Geistlich Pharma AG, Wolhusen, Switzerland) mixed with polynucleotide and hyaluronic acid-based gel (Regenfast®). The alveolus will be sealed with a porcine collagen membrane (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switzerland).
  Interventions: Procedure: Alveolar ridge preservation using DBBM + Regenfast + collagen matrix

INTERVENTIONS:
Procedure: Alveolar ridge preservation using DBBM + Regenfast + collagen matrix — Post extraction sites be filled up to the level of the highest point of the alveolar bone crest using particulate DBBM xenograft (Bio-Oss, Geistlich Pharma AG, Wolhusen, Switzerland) mixed with polynucleotide and hyaluronic acid-based gel (Regenfast®). The alveolus will be sealed with a porcine collagen membrane (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switzerland) and secured with 4-6 simple interrupted sutures (Resolon 6-0, Resorba Medical GmbH, Nuremberg, Germany).
  Arms: DBBM + Regenfast + collagen matrix
Procedure: Alveolar ridge preservation using DBBM + collagen matrix — Post extraction sites be filled up to the level of the highest point of the alveolar bone crest using particulate DBBM xenograft (Bio-Oss, Geistlich Pharma AG, Wolhusen, Switzerland). The alveolus will be sealed with a porcine collagen membrane (Mucograft Seal, Geistlich Pharma AG, Wolhusen, Switzerland) and secured with 4-6 simple interrupted sutures (Resolon 6-0, Resorba Medical GmbH, Nuremberg, Germany).
  Arms: DBBM + collagen matrix

SUMMARY:
Alveolar ridge resorption after tooth extraction is a physiological process that continues throughout the patient's life due to the loss of the periodontal ligament and lack of mechanical stimulation. Alveolar ridge preservation (ARP) techniques aim to minimize dimensional changes in the ridge after tooth extraction. These techniques involve grafting the socket to fill the bed and/or sealing it with a biomaterial. Currently, there is a polynucleotide and hyaluronic acid-based gel (Regenfast®) on the market that has proven useful in treating residual periodontal defects. Hyaluronic acid-based gels also appear to enhance the regenerative potential of critical bone defects in both in-vitro studies on rats and clinical studies. Therefore, this study aims to evaluate the clinical and histological effects of polynucleotide and hyaluronic acid-based gel in alveolar preservation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) who need the extraction of a single non-molar tooth in the mandible or maxilla.
* ASA I or II
* Intact post-extraction socket or with only one wall dehiscence (buccal or lingual) of no more than 50% of the socket.
* The treatment plan must include the replacement of the tooth to be extracted by placing an implant and an implant-supported prosthesis.

Exclusion Criteria:

* Mandibular incisors and molars.
* Acute infection associated with the tooth that needs to be extracted.
* Uncontrolled systemic disease.
* Pregnant patient.
* Patient under treatment with antiresorptives drugs (bisphosphonates or Receptor Activator of Nuclear Factor Kappa-B Ligand (i.e., Denosumab)) or antiangiogenics.
* Smokers (>10 cigarettes a day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric results | 3 months
  After 3 months of the ARP, A trephine with an internal diameter of 2.5 mm and a maximum length of 15 mm will be used to extract a bone core for histological analysis. Histological analyses will be performed on the entire sample area by calibrated and blinded examiners using open-source software (ImageJ, NIH). The areas of mineralized tissue and remaining xenograft material will be quantified based on their appearance and expressed as a percentage of the total area. The remaining area in the sample will be classified as non-mineralized tissue.

SECONDARY OUTCOMES:
Visual evaluation of socket healing. | At 1 week and 12 weeks
  Clinician will evaluate the healing of the socket based on a Healing index described by Avila-Ortiz, et al., 2018
Implant insertion torque | 3 months
  Implant insertion torque measured in N·cm
Need for additional bone regeneration for implant placement | 3 months
  Evaluation of the feasibility to place dental implant without needing additional bone regeneration
Dimensional changes | Measurement at the day of the ARP and 3 months
  Changes in the horizontal and vertical dimensions of the alveolar ridge after the ARP
Postoperative pain | During the first 7 postoperative days after ARP.
  Visual Analog scale.
Analgesic medication consumption | During the first 7 postoperative days after ARP.
  Record of analgesics and anti-inflammatory drugs used
Oral health related quality of life | At the day of the ARP and 7 days postoperative
  Evaluation of the quality of life of the patient after an ARP procedure by means of the validated questionnaire OHIP-14

CONTACTS AND LOCATIONS:
Overall Officials: Adria Jorba Garcia, DDS, MS, Principal Investigator — University of Barcelona; Javier Bara-Casaus, MD, PhD, Study Chair — University of Barcelona
Locations (1):
- Faculty of medicine and health sceince, University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Pilloni A, Rojas MA, Trezza C, Carere M, De Filippis A, Marsala RL, Marini L. Clinical effects of the adjunctive use of polynucleotide and hyaluronic acid-based gel in the subgingival re-instrumentation of residual periodontal pockets: A randomized, split-mouth clinical trial. J Periodontol. 2023 Mar;94(3):354-363. doi: 10.1002/JPER.22-0225. Epub 2022 Nov 23. PMID 36189651
- [Background] de Brito Bezerra B, Mendes Brazao MA, de Campos ML, Casati MZ, Sallum EA, Sallum AW. Association of hyaluronic acid with a collagen scaffold may improve bone healing in critical-size bone defects. Clin Oral Implants Res. 2012 Aug;23(8):938-42. doi: 10.1111/j.1600-0501.2011.02234.x. Epub 2011 Jun 21. PMID 21689163
- [Background] Cairo F, Cavalcanti R, Barbato L, Nieri M, Castelluzzo W, di Martino M, Pilloni A. Polynucleotides and Hyaluronic Acid (PN-HA) Mixture With or Without Deproteinized Bovine Bone Mineral as a Novel Approach for the Treatment of Deep Infrabony Defects: A Retrospective Case Series. Int J Periodontics Restorative Dent. 2025 Mar 6;45(2):153-163. doi: 10.11607/prd.7065. PMID 38363180